CLINICAL TRIAL: NCT05019482
Title: Effects of an Intervention Among University Student to Promote Physical Activity and Reduce the Sedentary Time During COVID-19 Pandemic
Brief Title: Intervention Program Among University Student to Promote Physical Activity and Reduce the Sedentary Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nimes (Other)
Responsible Party: Principal Investigator, aurelie goncalves, Associate professor, University of Nimes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNimes.2
Record Dates: First submitted 2021-07-22; First posted 2021-08-24 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Physical Activity; Sedentary Behavior; Young Adults; Student
Keywords: Physical Activity; Sedentary Behavior; student
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: During the, baseline assessments were carried out in two groups (Experimental group, control group): measures of PA, ST, anthropometric data, sleep, physical condition and psychological variables (motivation, body appreciation, perceived control, well-being, …) These assessments were performed in October 2021 (First Time - T1) and December 2021 (Second time - T2).
  During the first academic semester, a university-based intervention to increase PA and reduce ST was realised in Experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- University-based 8-weeks intervention to promote Physical Activity (PA) (Experimental): Experimental group: 8-weeks program of Physical Activity constructed by users during a design-based innovative workshops before the beginning of the interventions .
  Interventions: Behavioral: University-based intervention to promote PA and reduce ST
- Control Group (No Intervention): Control group: No intervention, only two measurement times

INTERVENTIONS:
Behavioral: University-based intervention to promote PA and reduce ST — This intervention was realized with all college student and involved:
  1. Design-based innovative workshops during the first week;
  2. 8-weeks program of Physical Activity constructed by users
  3. Information session focusing on the promotion of active behaviors
  4. Feedback provided to the users with an individualized report
  Arms: University-based 8-weeks intervention to promote Physical Activity (PA)

SUMMARY:
Since the beginning of the COVID-19 pandemic, university students have faced many challenges and without any preparation. Studies conducted during the first lockdown show an increase in unhealthy lifestyles.

This study will be proposed to students from University of Nimes an 8-week physical activity program. Two groups will be constituted: the first will benefit from of innovative physical activity program on the base of the co-construction with users (Experimental Group), another that will not benefit from any intervention (Control Group). Investigators plan to include approximately 90 university students, 45 in each group.

The main goal of the study is to propose innovative program to promote PA (Physical Activity) and reduce ST (Sedentary Time) of young adults aged over 18 from university of Nîmes. The levels of PA and ST of the experimental group will be compared to a control group with the realization of pre and post intervention measures.

DETAILED DESCRIPTION:
In March 2020, the World Health Organization declared the coronavirus disease 2019 (COVID-19) as a global pandemic. In France, all universities have been closed on 16th March 2020. In September 2020, face-to-face teaching restarted in French universities, but with new constraints (e.g., reducing number of students in classrooms, wearing masks) and significant changes in teachings (e.g., distance and/or hybrid education). In October 2020, several French universities closed down again due to significant contamination among students. Finally, on 30th October 2020, the French government imposed a second lockdown and all universities have been closed. It is only in February 2021 that face-to-face teaching started again in French universities (within the limit of 50% of the universities' capacity and 20% of the teachings). Since the beginning of the pandemic, university students have faced many challenges and without any preparation.

Even before the pandemic, university students were identified as a population with unhealthy lifestyles and habits, notably reflected in high levels of sedentary behavior, low levels of physical activity and unhealthy diet. Studies conducted during the first lockdown have shown an increase in unhealthy lifestyles;

The deleterious effects of the pandemic on students' health are now evident. However, some areas of research are still under-explored.

1. The majority of research is largely descriptive and do not identify the factors involved in the deterioration of health
2. To date, no interventional studies have been conducted to prevent the deterioration of students' health.

Investigators expect a 9-week intervention. During the first week, a workshop of the co-construction with the users will be realized in order to remove the barriers to the practice of a physical activity. The aim of co-construction with users is to obtain better adherence to program, based on needs and not decided from above. Then, a group information session focusing on the promotion of active behaviors will be organize, and physical activities (moderate to vigorous) will be proposed for 8 weeks, twice a week.

The main goal of the study is to propose innovative program to promote PA (Physical Activity) and reduce ST (Sedentary Time) of young adults aged over 18 from university of Nîmes. The levels of PA and ST of the experimental group will be compared to a control group with the realization of pre and post intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* Students at the University of Nimes

Exclusion Criteria:

* Physical diseases that prevent PA practice
* Depending on the evolution of sanitary conditions and governmental instructions in relation to COVID-19, the absence of a negative PCR test or vaccination may be a criterion for exclusion
* not to be a student of the University of Nîmes
* not signing the consent form to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Change in level of physical activity (PA) | Baseline and post-intervention (8-week)
  Physical activity, is measured with tri-axis accelerometers of the brand Actigraph model GT3X (Actilife, Pensacola, FL, USA). Data is collected every 10 seconds during 5 consecutive whole days. It is the most feasible and precise method for the purpose.
Sedentary Time (ST) | Baseline and post-intervention (8-week)
  Sedentary Time (ST), is measured with tri-axis accelerometers of the brand Actigraph model GT3X (Actilife, Pensacola, FL, USA). Data is collected every 10 seconds during 5 consecutive whole days. It is the most feasible and precise method for the purpose.

SECONDARY OUTCOMES:
Change in body fat | Baseline and post-intervention (8-week)
  Body fat composition will be assessed trought a Bioelectrical Impedance Analysis method using a Tanita 780 MA-S Body Composition Analyser/Scale.
  Body fat is expressed as body fat mass (kg) and body fat percentage (%).
Change in body muscle | Baseline and post-intervention (8-week)
  Body muscle composition will be assessed trought a Bioelectrical Impedance Analysis method using a Tanita 780 MA-S Body Composition Analyser/Scale.
  Body muscle is expressed as body muscle mass (kg) and body muscle percentage (%).
Change in body water | Baseline and post-intervention (8-week)
  Body water composition will be assessed trought a Bioelectrical Impedance Analysis method using a Tanita 780 MA-S Body Composition Analyser/Scale.
  Body water is expressed as body water mass (kg) and body water percentage (%).
Change in visceral fat rating | Baseline and post-intervention (8-week)
  Visceral fat rating will be assessed trought a Bioelectrical Impedance Analysis method using a Tanita 780 MA-S Body Composition Analyser/Scale.
  Visceral fat rating is expressed on a scale from 1 to 60. A score between 1 and 12 is considering as healthy and a score between 12 to 60 is considering as excessive.
Body Mass Index (BMI) | Baseline and post-intervention (8-week)
  Height and weight will be measured by study staff at the baseline visit using a stadiometer (collecting height measures twice and reporting the average) and a calibrated scale TANITA 780 MA-S (light clothing, street shoes removed).
  BMI will be calculated as weight in kilograms divided by height in squared centimeters. Weight will be re-measured at 8 week.
Changes in Physical Fitness : cardiovascular fitness | Baseline and post-intervention (8-week)
  Participants complete a YMCA 3-minute step test for cardiovascular fitness (assessment of resting heart rate and recovery heart rate)
Changes in Physical Fitness: flexibility | Baseline and post-intervention (8-week)
  Participants complete a sit-and-reach test for flexibility
Changes in Physical Fitness: strength upper limb. | Baseline and post-intervention (8-week)
  Participants complete a grip strength test for strength of upper limb.
  Hand-grip strength measurement is made with a hydraulic hand-grip dynamometer. Hand-grip strength measurement is performed for the dominant hand when the elbow is close to the body, 90 degrees of flexion, and the wrist is in a neutral position. The measurement is repeated 3 times and the maximum value is recorded in kg. The dominant hand is determined by asking the participants with which hand they write.
Changes in Physical Fitness: strength lower limb. | Baseline and post-intervention (8-week)
  Participants complete a muscular lower limb strength test measured with the dynamometric chair LegControl V2.
Quality of sleep, defined by number and duration of awakenings, and longest sustained sleep period for the study interval. | Baseline and post-intervention (8-week)
  These data were measured by the Actigraph model GT3X (Actilife, Pensacola, FL, USA)and summarized as percentage of time spent sleeping, or sleep efficiency. Data is collected every 10 seconds during 5 consecutive whole days.

OTHER OUTCOMES:
Changes in Physical Activity as measured by the International Physical Activity - Short Form (IPAQ-SF) | Baseline and post-intervention (8-week)
  Subjective physical activity and sitting time over the last 7 days are measured.
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in motivation | Baseline and post-intervention (8-week)
  Motivation is assessed with he motivation scale towards health-oriented physical activity in french.
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in sleep quality (PSQI) | Baseline and post-intervention (8-week)
  Assessment of sleep quality is measured with the French adaptation of Pittsburgh Sleep Quality Index (PSQI). It is a simple tool which assess the sleep quality over one month period. It included seven components with a global PSQI score > 5 is indicative of poor sleep quality
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in body image (BAS-2) | Baseline and post-intervention (8-week)
  Assessment of body image measured with the Body Appreciation Scale-2 (BAS-2). The scale comprises 10 items rated on a 5-point scale, ranging from 1 (Never) to 5 (Always), with higher total scoring indicating more positive body appreciation.
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in eating behaviors (EAT-26) | Baseline and post-intervention (8-week)
  Assessment of eating behaviour measured with the eating Attitudes Test (EAT-26).
  The EAT-26 is a self-administered questionnaire that reveals abnormal eating behaviors. It consists of 26 items with six components scored from 0 to 3 (Zero: "Never," "Rarely," and "Sometimes"; 1: "Often"; 2: "Very often"; and 3: "Always"). The total score range from 0 to 78, and a score ≥ 20 is considered to represent abnormal eating attitudes or behaviors
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in Anxiety and depressive symptoms (HADS) | Baseline and post-intervention (8-week)
  Assessment of anxiety and depressive symptoms measured with the Hospital Anxiety and Depression Scale (HADS).
  These symptoms are assessed using a French version of the HADS. This 14-item self-report questionnaire assesses anxiety symptoms and depressive symptoms (7 items for each dimension) with labels varying from one item to the next. Scores range from 0 to 21 for each dimension, with higher scores reflecting higher levels of anxiety or depressive symptoms.
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in social support (SPS-10) | Baseline and post-intervention (8-week)
  Assessment of social support measured with the french validation of the Social Provisions Scale-10 item
  The 10 items are rated on a 4-point Likert scale ranging from 1 ("strongly disagree") to 4 ("Strongly in agreement").
  This self-report scale capturing five dimensions of social support (two items per dimension of support): emotional support or attachment (e.g., "I feel a strong emotional bond with at least one other person"), social integration (e.g., "there are people who enjoy the same social activities I do"), reassurance of worth (e.g., "there are people who admire my talents and skills"), tangible help (e.g., "there are people I can count on to help me when I really need it"), and orientation (e.g., "there is someone with whom I can discuss important decisions about my life").
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in well-being | Baseline and post-intervention (8-week)
  Assessment of well-being is evaluated with the French validation of the psychological Well-Being Scale. The 18 items are rated on a 6-point Likert scale ranging from 1 ("Disagreement") to 6 ("Agreement"). This self-report scale capturing six components of weel-being (three items per components): autonomy, control of the environment, personal development, positive relationships, giving meaning to life and self-acceptance.
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in perceived fatigue (MFI-20) | Baseline and post-intervention (8-week)
  Assessment of perceived fatigue is evaluated with the French validation of the Multidimensional Fatigue Inventory (MFI-20)
  A self-report instrument of five dimensions of fatigue. General fatigue, physical fatigue, mental fatigue, reduced activity and reduced motivation.
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Changes in perceived control (PSMS) | Baseline and post-intervention (8-week)
  Assessment of well-being is evaluated with the French validation of the the Pearlin Self-Mastery Scale Perceived control with scores range up to 28, higher scores = higher mastery
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Situational factors | Baseline and post-intervention (8-week)
  Investigators considered six situational factors:
  1. the extent to which participants felt that lockdown was compromising their future job prospects (scale ranging from 0 to 100)
  2. the extent to which university studies were essential to participants (scale ranging from 0 to 100)
  3. the presence or absence of COVID symptoms (dichotomous answer: Yes or No)
  4. the presence or absence of COVID symptoms in their relatives (dichotomous answer: Yes or No)
  5. participants' level of concern about their health owing to the COVID-19 crisis (scale ranging from 0 to 100)
  6. participants' level of concern about their relatives' health owing to the COVID-19 crisis (scale ranging from 0 to 100).
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).
Socio-demographic factors | Baseline
  Investigators considered four socio-demographic factors:
  1. Age
  2. Gender
  3. Level of education
  4. Field of study
  Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).

CONTACTS AND LOCATIONS:
Overall Officials: ELODIE CHARBONNIER, PhD, Study Director — UNIVERSITE DE NIMES - UPR APSY-v
Locations (1):
- Universite de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charbonnier E, Tremoliere B, Baussard L, Goncalves A, Lespiau F, Philippe AG, Le Vigouroux S. Effects of an online self-help intervention on university students' mental health during COVID-19: A non-randomized controlled pilot study. Comput Hum Behav Rep. 2022 Mar;5:100175. doi: 10.1016/j.chbr.2022.100175. Epub 2022 Feb 10. PMID 35169655
- [Background] Charbonnier, E., Le Vigouroux, S., & Goncalves, A. (2021). Etudiants en temps de confinement et au-delà. La Presse Médicale Formation. https://doi.org/10.1016/j.lpmfor.2021.06.011
- [Background] Ait-Aoudia M, Levy PP, Bui E, Insana S, de Fouchier C, Germain A, Jehel L. Validation of the French version of the Pittsburgh Sleep Quality Index Addendum for posttraumatic stress disorder. Eur J Psychotraumatol. 2013 Sep 12;4. doi: 10.3402/ejpt.v4i0.19298. eCollection 2013. PMID 24044071
- [Background] Boiche J, Gourlan M, Trouilloud D, Sarrazin P. Development and validation of the 'Echelle de Motivation envers l'Activite Physique en contexte de Sante': A motivation scale towards health-oriented physical activity in French. J Health Psychol. 2019 Mar;24(3):386-396. doi: 10.1177/1359105316676626. Epub 2016 Nov 21. PMID 27872385
- [Background] Lepine JP, Godchau M, Brun P. Anxiety and depression in inpatients. Lancet. 1985 Dec 21-28;2(8469-70):1425-6. doi: 10.1016/s0140-6736(85)92589-9. No abstract available. PMID 2867417
- [Background] Castro O, Bennie J, Vergeer I, Bosselut G, Biddle SJH. Correlates of sedentary behaviour in university students: A systematic review. Prev Med. 2018 Nov;116:194-202. doi: 10.1016/j.ypmed.2018.09.016. Epub 2018 Sep 25. PMID 30266213
- [Background] Castro O, Bennie J, Vergeer I, Bosselut G, Biddle SJH. How Sedentary Are University Students? A Systematic Review and Meta-Analysis. Prev Sci. 2020 Apr;21(3):332-343. doi: 10.1007/s11121-020-01093-8. PMID 31975312
- [Background] Deliens T, Van Crombruggen R, Verbruggen S, De Bourdeaudhuij I, Deforche B, Clarys P. Dietary interventions among university students: A systematic review. Appetite. 2016 Oct 1;105:14-26. doi: 10.1016/j.appet.2016.05.003. Epub 2016 May 13. PMID 27181201
- [Background] Galle F, Sabella EA, Ferracuti S, De Giglio O, Caggiano G, Protano C, Valeriani F, Parisi EA, Valerio G, Liguori G, Montagna MT, Romano Spica V, Da Molin G, Orsi GB, Napoli C. Sedentary Behaviors and Physical Activity of Italian Undergraduate Students during Lockdown at the Time of CoViD-19 Pandemic. Int J Environ Res Public Health. 2020 Aug 25;17(17):6171. doi: 10.3390/ijerph17176171. PMID 32854414
- [Background] Huckins JF, daSilva AW, Wang W, Hedlund E, Rogers C, Nepal SK, Wu J, Obuchi M, Murphy EI, Meyer ML, Wagner DD, Holtzheimer PE, Campbell AT. Mental Health and Behavior of College Students During the Early Phases of the COVID-19 Pandemic: Longitudinal Smartphone and Ecological Momentary Assessment Study. J Med Internet Res. 2020 Jun 17;22(6):e20185. doi: 10.2196/20185. PMID 32519963
- [Background] Kertechian S, Swami V. An examination of the factor structure and sex invariance of a French translation of the Body Appreciation Scale-2 in university students. Body Image. 2017 Jun;21:26-29. doi: 10.1016/j.bodyim.2017.02.005. Epub 2017 Mar 6. PMID 28260632
- [Background] Rodriguez-Larrad A, Manas A, Labayen I, Gonzalez-Gross M, Espin A, Aznar S, Serrano-Sanchez JA, Vera-Garcia FJ, Gonzalez-Lamuno D, Ara I, Carrasco-Paez L, Castro-Pinero J, Gomez-Cabrera MC, Marquez S, Tur JA, Gusi N, Benito PJ, Moliner-Urdiales D, Ruiz JR, Ortega FB, Jimenez-Pavon D, Casajus JA, Irazusta J. Impact of COVID-19 Confinement on Physical Activity and Sedentary Behaviour in Spanish University Students: Role of Gender. Int J Environ Res Public Health. 2021 Jan 6;18(2):369. doi: 10.3390/ijerph18020369. PMID 33418907
- [Background] Caron J. [A validation of the Social Provisions Scale: the SPS-10 items]. Sante Ment Que. 2013 Spring;38(1):297-318. doi: 10.7202/1019198ar. French. PMID 24337002
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Result] Le Vigouroux S, Goncalves A, Charbonnier E. The Psychological Vulnerability of French University Students to the COVID-19 Confinement. Health Educ Behav. 2021 Apr;48(2):123-131. doi: 10.1177/1090198120987128. Epub 2021 Jan 20. PMID 33472453
- [Derived] Goncalves A, Bernal C, Korchi K, Nogrette M, Deshayes M, Philippe AG, Gisclard B, Charbonnier E. Promoting Physical Activity Among University Students During the COVID-19 Pandemic: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 13;11(6):e36429. doi: 10.2196/36429. PMID 35700019